CLINICAL TRIAL: NCT00284141
Title: A Multicenter, Open-label, Single-arm, Two-stage Study of the Efficacy and Safety of AVE0005 (VEGF Trap) Administered Intravenously Every 2 Weeks in Patients With Platinum- and Erlotinib-resistant Locally Advanced or Metastatic Non-small-cell Lung Adenocarcinoma
Brief Title: Study of AVE0005 (VEGF Trap) in Locally Advanced or Metastatic Platinum- and Erlotinib- Resistant Non-small-cell-lung Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD6123; AVE0005B/2001
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2011-07

CONDITIONS: Pulmonary Diseases; Neoplasms, Lung
Keywords: lung; cancer; non-small-cell lung cancer; metastatic; carcinoma; lung neoplasm; lung diseases; angiogenesis; anti-angiogenesis; anti-angiogenesis inhibitors; cancer and other neoplasms; respiratory tract; (lung and bronchial) diseases
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms; Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis; Carcinoma; Disease | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- aflibercept 4.0 mg/kg (Experimental): Participants with metastatic non-small-cell lung adenocarcinoma administered 4.0 mg/kg Aflibercept every 2 weeks until a study withdrawal criterion was met.
  Interventions: Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®)

INTERVENTIONS:
Drug: Aflibercept (ziv-aflibercept, AVE0005, VEGF trap, ZALTRAP®) — Aflibercept 4.0 mg/kg administered intravenously (IV) over a period of at least 1 hour once every 2 weeks.
  Aflibercept could be reduced by 1 dose level (to 3.0 mg/kg) or 2 dose levels (to 2.0 mg/kg) in case of uncontrolled hypertension or urinary protein >3.5 g/24 hours. Intrapatient dose escalation was not to be permitted. Participants requiring more than 2 dose level reductions would be withdrawn from study treatment.

SUMMARY:
This study evaluated the efficacy and safety of aflibercept in the treatment of participants with advanced chemoresistant non-small cell lung adenocarcinoma (NSCLA).

Primary objective:

* To determine the overall objective response rate (ORR) of AVE0005 (ziv-aflibercept, aflibercept, VEGF trap, ZALTRAP®) 4.0 mg/kg intravenously (IV) every 2 weeks in participants with platinum- and erlotinib-resistant, locally advanced or metastatic NSCLA.

Secondary objective:

* To assess duration of response (DR), progression-free survival (PFS), and overall survival (OS) in this participant population
* To evaluate the safety profile of IV AVE0005 (ziv-aflibercept, aflibercept, VEGF trap, ZALTRAP®).

This study employed an Independent Review Committee (IRC) for radiological tumor assessments. For all tumor assessment-related efficacy variables, two analyses were performed: the primary analysis was based on Independent Review Committee (IRC) reviewed data and the secondary analysis was based on Investigator evaluation.

In addition, both Response Evaluation Criteria In Solid Tumors (RECIST) and Modified Response Evaluation Criteria In Solid Tumors (mRECIST) were used to assess tumors. Where as RECIST criteria only consider the longest diameter of the tumors for calculations pertaining to changes in tumor size, mRECIST assessments also account for the differences in the cavities of lesions observed in non-small-cell lung cancer (NSCLC). Responses based on RECIST and mRECIST are reported.

DETAILED DESCRIPTION:
The study included :

* A screening phase up to 21 days followed by registration
* Treatment initiation within 5 working days of registration
* A treatment phase with 14-day study treatment cycles until a study withdrawal criterion was met or up to the clinical database cut-off date (18 July 2008)
* A follow-up phase - up to 60 days after end of treatment

Withdrawal criteria that led to treatment discontinuation were:

* The participant or their legally authorized representative requested to withdraw
* In the investigator's opinion, continuation of the study would be detrimental to the participant's well being, due to reasons such as disease progression, unacceptable toxicity, noncompliance, or logistical considerations.
* A specific request by the Sponsor
* Participant had intercurrent illness that prevented further administration of study treatment
* Participant had more than 2 aflibercept dose reductions
* Participant had arterial thromboembolic events, including cerebrovascular accidents, myocardial infarctions, transient ischemic attacks, new onset or worsening of pre-existing angina
* Participant had radiographic evidence of intestinal obstruction (e.g., dilated loops of bowel accompanied by air-fluid levels) or gastrointestinal perforation (e.g., presence of extraluminal gas) requiring surgical intervention
* Participant was lost to follow-up

After discontinuing treatment, participants remained on the study until the last post-treatment visit or until recovery of drug related toxicities, whichever was later.

ELIGIBILITY:
Participants who met the following criteria were eligible for the study.

Inclusion Criteria:

* Histologically confirmed non-small-cell lung adenocarcinoma that is locally advanced or metastatic
* Prior treatment with at least 2 cancer drug regimens in the advanced disease setting
* Platinum- and erlotinib-resistant disease defined by relapse or progression during or after treatment
* Measurable disease by RECIST criteria
* ECOG Performance status less than or equal to 2
* Resolution of any toxic effects of prior therapy
* Adequate organ and bone marrow function
* Female patients must be post-menopausal, surgically sterile or using effective contraception
* Willing and able to comply with study procedures and sign informed consent

Exclusion Criteria:

* Diagnosis of squamous-cell lung cancer or any second malignancy within the last 5 years (except for adequately treated basal cell or squamous cell skin cancer or in situ carcinoma of the cervix uteri)
* Prior treatment with a VEGF or VEGF receptor inhibitor with the exception of bevacizumab (Avastin-TM)
* Anticipation of a need for major surgical procedure
* Treatment with chemotherapy, radiotherapy, surgery, blood products, or an investigational agent within 3 weeks (6 weeks for nitrosoureas, mitomycin C, immunotherapy, or cytokine therapy) of study enrollment
* Uncontrolled hypertension
* Any severe or acute medical or psychiatric problem within the past 6 months requiring further investigation or that may cause undue risk for the patient's safety
* History of brain metastases, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease
* Active infection or on antiretroviral therapy for HIV disease
* Pregnant or breast-feeding

The above information is not intended to contain all considerations relevant to potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (3):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Paris, France

REFERENCES:
- [Result] Leighl NB, Raez LE, Besse B, Rosen PJ, Barlesi F, Massarelli E, Gabrail N, Hart LL, Albain KS, Berkowitz L, Melnyk O, Shepherd FA, Sternas L, Ackerman J, Shun Z, Miller VA, Herbst RS. A multicenter, phase 2 study of vascular endothelial growth factor trap (Aflibercept) in platinum- and erlotinib-resistant adenocarcinoma of the lung. J Thorac Oncol. 2010 Jul;5(7):1054-9. doi: 10.1097/jto.0b013e3181e2f7fb. PMID 20593550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 98 participants were registered into the study, of whom, 96 were exposed to study treatment.
Groups:
- Aflibercept 4.0 mg/kg: Participants with metastatic non-small-cell lung adenocarcinoma administered 4.0 mg/kg Aflibercept intravenously every 2 weeks until a study withdrawal criterion was met.
Period: Overall Study
Arm/Group | Aflibercept 4.0 mg/kg
Started | 98
TREATED | 96 (Participants received at least part of one dose of Aflibercept.)
ONGOING TREATMENT | 2 (Participants were still on study treatment at the clinical database cut-off date.)
Completed | 0 (Participants met treatment discontinuation criteria or were still ongoing treatment.)
Not Completed | 98
Not completed — Disease Progression / Lack of efficacy | 51
Not completed — Adverse Event | 19
Not completed — Participant's request | 9
Not completed — Symptomatic / Clinical Progression | 11
Not completed — Clinical deterioration / death | 2
Not completed — General decline | 1
Not completed — Pneumonia | 1
Not completed — Did not take study medication | 2
Not completed — Ongoing treatment | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 98
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 40
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 79
  Black | 3
  Asian, Oriental | 5
  Unknown or Not Reported | 11

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response (OR) Based Upon Modified Response Evaluation Criteria in Solid Tumors (RECIST) Assessed by the Independent Review Committee (IRC).
Description: OR was either complete response (CR) or partial response (PR) based on RECIST or modified RECIST. CR was the disappearance of all target/nor-target lesions; and PR was at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, with reference to the baseline sum LD (According to modified RECIST, to calculate LD for cavitated lesions, the longest cavitation diameters were subtracted from the LD of cavitated target lesions).
  Assessments were made by the IRC, and confirmed by repeat tumor imaging 4-6 weeks after documentation of the initial response.
Time Frame: up to 2.5 years from initial treatment
Population: Simon's cohort: The first 84 evaluable participants, based on Simon's two-stage study design that required 84 evaluable participants to maintain a targeted 90% power.
Measure: Number; unit: Participants
Groups:
- Aflibercept 4.0 mg/kg Arm Assessed by Modified RECIST: Participants with metastatic non-small-cell lung adenocarcinoma administered 4.0 mg/kg Aflibercept intravenously every 2 weeks assessed by RECIST criteria.
- Aflibercept 4.0 mg/kg Arm Assessed by RECIST: Participants with metastatic non-small-cell lung adenocarcinoma administered 4.0 mg/kg Aflibercept intravenously every 2 weeks assessed by modified RECIST criteria.
Arm/Group | Aflibercept 4.0 mg/kg Arm Assessed by Modified RECIST | Aflibercept 4.0 mg/kg Arm Assessed by RECIST
Number analyzed (Participants) | 84 | 84
Participants | 0 | 0

2. Secondary Outcome: Duration of Response (DR)
Description: DR was the time interval from the first complete response (CR) or partial response (PR) to the date of tumor progression or death from any cause, whichever was earlier. The duration of response was calculated only for those participants who achieved CR or PR.
Time Frame: up to 2.5 years from initial treatment
Population: No modified RECIST responses, as confirmed by the IRC review, were observed. Only 2 responders were reported by the Investigators. Therefore, the analyses for duration of response was not performed.
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival (PFS) Time Assessed by the Independent Review Committee (IRC)
Description: PFS time was interval from the date of registration to the date of tumor progression (by RECIST or modified RECIST), or death from any cause, whichever was earlier. Median PFS time was estimated from Kaplan-Meier Plots.
  Progression was at least a 20% increase in the sum of the longest diameter (LD) of tumors, compared to smallest sum LD recorded since treatment started, or the appearance of one or more new tumors.
  If a participant did not progress or die, the date was censored to the date of last valid tumor assessment or the date of data cut-off, whichever was earlier.
Time Frame: up to 2.5 years from initial treatment
Population: All registered participants. 18 participants were censored.
Measure: Median (95% Confidence Interval); unit: weeks
Units Other Than Participants: Participants with PFS Events
Arm/Group | Aflibercept 4.0 mg/kg Arm Assessed by Modified RECIST | Aflibercept 4.0 mg/kg Arm Assessed by RECIST
Number analyzed (Participants) | 98 | 98
Number analyzed (Participants with PFS Events) | 80 | 80
weeks | 11.3 [9.3 to 16.1] | 11.3 [9.3 to 16.1]

4. Secondary Outcome: Progression-free Survival (PFS) Time Assessed by the Investigator
Description: PFS time was interval from the date of registration to the date of tumor progression (by RECIST or modified RECIST), or death from any cause, whichever was earlier. If a participant did not progress or die, the date was censored to the date of last valid tumor assessment or the date of data cut-off, whichever was earlier. Median PFS time was estimated from Kaplan-Meier Plots.
  Progression was at least a 20% increase in the sum of the longest diameter (LD) of tumors, compared to smallest sum LD recorded since treatment started, or the appearance of one or more new tumors.
Time Frame: up to 2.5 years from initial treatment
Population: All registered participants. 17 participants were censored.
Measure: Median (95% Confidence Interval); unit: weeks
Units Other Than Participants: Participants with PFS Events
Arm/Group | Aflibercept 4.0 mg/kg Arm Assessed by Modified RECIST | Aflibercept 4.0 mg/kg Arm Assessed by RECIST
Number analyzed (Participants) | 98 | 98
Number analyzed (Participants with PFS Events) | 81 | 81
weeks | 12.0 [10.0 to 16.0] | 11.9 [9.7 to 14.7]

5. Secondary Outcome: Overall Survival (OS)
Description: OS was the time interval between registration to the date of death from any cause. The median time for OS was estimated from Kaplan-Meier Plots.
  A participant was to be censored for the OS analysis if the participant was alive by the study cut-off date. The censoring date was either the date that the participant was last known to be alive or the date of study cut-off, whichever came earlier.
Time Frame: up to 2.5 years from initial treatment
Population: All registered participants. 38 participants were censored for OS.
Measure: Median (95% Confidence Interval); unit: months
Units Other Than Participants: Participant with OS Event (death)
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 98
Number analyzed (Participant with OS Event (death)) | 60
months | 26.9 [21.0 to 49.3]

6. Secondary Outcome: Heath-related Quality of Life (QOL) Measured Via the Lung Cancer Subscale
Description: HRQL was assessed with the Functional Assessment of Cancer Therapy-Lung Cancer Subscale (FACT-LCS) questionnaire, which was completed by the participants on Day 1 of Cycle 1 only (for baseline value), then on Day 14 of each even-numbered cycle to evaluate the participants symptoms.
  The questionnaire scored 7 symptoms: shortness of breath, weight loss, clarity in thinking, coughing, appetite, chest tightness, ease of breathing, on a 0-4 scale. The total FACT-LCS score ranged from 0-28 (where 28 was related to the worst outcome). To calculate a change, the baseline score was subtracted from the score obtained after treatment. A negative value implied an improvement in HRQL.
Time Frame: Baseline to 2.5 years
Population: All registered participants with available questionnaires at the timepoint assessed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 83
score on a scale
  Baseline FACT-LCS Score (N=83) | 19.9 (3.9)
  Change from baseline at Cycle 2 (N=58) | -1.5 (3.6)
  Change from baseline at Cycle 4 (N=41) | -1.9 (4.7)
  Change from baseline at Cycle 6 (N=25) | -1.0 (5.0)
  Change from baseline at Cycle 8 (N=13) | -1.4 (4.7)
  Change from baseline at Cycle 10 (N=10) | -1.7 (6.9)
  Change from baseline to last assessment (N=70) | -3.3 (5.2)

7. Secondary Outcome: Overall Safety - Number of Participants With Adverse Events
Description: All AEs regardless of seriousness or relationship to study treatment, spanning from the first administration of study treatment until 60 days after the last administration of study treatment, were recorded, and followed until resolution or stabilization. The number of participants with all treatment emergent adverse events (TEAE), serious adverse events (SAE), TEAE leading to death, and TEAE leading to permanent treatment discontinuation are reported.
Time Frame: up to 60+/-5 days after treatment discontinuation, or or until TEAE was resolved or stabilized (Collected till 18 July 2008)
Population: All participants who received at least part of 1 dose of study treatment.
Measure: Number; unit: participants
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 96
participants
  With any TEAE | 96
  With any Serious TEAE | 47
  With any TEAE leading to Death | 16
  with any TEAE leading to Treatment discontinuation | 19

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Participants with abnormal laboratory results for
  * Liver and renal function (Alkaline phosphatase, Alanine aminotransferase [ALT], aspartate aminotransferase [AST], Creatinine, Hyperbilirubinemia),
  * Electrolytes (Hypercalcemia, Hypocalcemia, Hypokalemia, Hypernatremia, Hyponatremia, Hypophosphatemia)
  * Metabolism (Hypoalbuminemia, Hyperglycemia, Hypoglycemia)
  * Hematology (Partial thromboplastin time, Anemia, Lymphopenia, Neutropenia, Thrombocytopenia, Leukopenia)
Time Frame: Up to 2.5 years
Population: All participants who received at least part of 1 dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 96
Participants
  LIVER AND RENAL FUNCTION- Alkaline Phosphatase | 39
  LIVER AND RENAL FUNCTION - ALT | 35
  LIVER AND RENAL FUNCTION - AST | 37
  LIVER AND RENAL FUNCTION - Creatinine | 15
  LIVER AND RENAL FUNCTION - Hyperbilirubinemia | 4
  ELECTROLYTES - Hypercalcemia | 6
  ELECTROLYTES - Hypocalcemia | 15
  ELECTROLYTES - Hyperkalemia | 24
  ELECTROLYTES - Hypokalemia | 10
  ELECTROLYTES - Hypernatremia | 5
  ELECTROLYTES - Hyponatremia | 41
  ELECTROLYTES - Hypophosphatemia (N=91) | 14
  METABOLISM - Hypoalbuminemia (N=91) | 44
  METABOLISM - Hyperglycemia | 81
  METABOLISM - Hypoglycemia | 10
  HEMATOLOGY - Partial thromboplastin time (N=81) | 30
  HEMATOLOGY - Anemia | 34
  HEMATOLOGY - Lymphopenia (N=84) | 60
  HEMATOLOGY - Neutropenia (N=78) | 4
  HEMATOLOGY - Thrombocytopenia | 11
  HEMATOLOGY - Leukopenia | 11

9. Secondary Outcome: Peak of Free Aflibercept (VEGF Trap)
Description: Plasma free aflibercept levels after the first aflibercept infusion were estimated by a validated direct measured by enzyme-linked immunosorbent assay (ELISA), with a limit of quantification (LOQ) of 15.6 ng/mL.
Time Frame: Day 1 of the first infusion of Aflibercept (cycle 1)
Population: All participants who received at least part of 1 dose of study treatment and had evaluable blood samples.
Measure: Mean (Standard Deviation); unit: micrograms/mL
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 47
micrograms/mL | 71.4 (31.8)

10. Secondary Outcome: Free and VEGF-bound Trough Aflibercept Concentrations (VEGF Trap)
Description: Median free and VEGF-bound trough concentrations were determined at the end of each cycle beyond Cycle 2 (Steady-state) for each participant.
  Plasma free aflibercept levels were estimated by a validated direct ELISA, with an LOQ of 15.6 ng/mL. Plasma VEGF-bound aflibercept levels were also estimated by a separate validated direct ELISA with an LOQ of 43.9 ng/mL.
  Mean ± SD (coefficient of variation [CV%]) values were estimated from the median values calculated for each participant.
Time Frame: At the end of each treatment cycle (up to 2.5 years)
Population: All participants who received at least part of 1 dose of study treatment and had evaluable blood samples on Day 1 of Cycle 3 for measurement of VEGF-bound aflibercept.
Measure: Mean (Standard Deviation); unit: micrograms/mL
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 61
micrograms/mL
  Trough free aflibercept concentration | 9.53 (6.28)
  Trough VEGF-bound aflibercept concentration | 3.48 (1.04)

11. Primary Outcome: Confirmed Objective Response Based Upon Modified Response Evaluation Criteria in Solid Tumors (RECIST) Assessed by the Investigator.
Description: OR was either complete response (CR) or partial response (PR) based on RECIST or modified RECIST. CR was the disappearance of all target/nor-target lesions; and PR was at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, with reference to the baseline sum LD (According to modified RECIST, to calculate LD for cavitated lesions, the longest cavitation diameters were subtracted from the LD of cavitated target lesions).
  Assessments were made by the Investigator, and confirmed by repeat tumor imaging 4-6 weeks after documentation of the initial response.
Time Frame: up to 2.5 years from initial treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Aflibercept 4.0 mg/kg Arm Assessed by Modified RECIST | Aflibercept 4.0 mg/kg Arm Assessed by RECIST
Number analyzed (Participants) | 84 | 84
participants
  Objective response (OR) | 2 | 2
  Complete response (CR) | 0 | 0
  Partial response (PR) | 2 | 2

12. Secondary Outcome: Number of Participants With Anti-drug Antibodies
Description: Anti-drug antibodies in a participant's serum sample were assayed with an anti-drug ELISA assay, with a lower limit of quantitation of 238.4 ng/mL for an undiluted human serum sample.
  Serum for anti-drug antibody analysis was collected pre-dose on every fourth cycle after Cycle 1 Day 1 (at 8 week intervals), at end of treatment (EOT), and during post-treatment follow-up 60 days after the last dose.
Time Frame: up to 2.5 years after initial treatment
Population: All participants who received at least part of 1 dose of study treatment and had evaluable blood samples.
Measure: Number; unit: participants
Arm/Group | Aflibercept 4.0 mg/kg
Number analyzed (Participants) | 80
participants | 0

ADVERSE EVENTS:
Time Frame: From treatment initiation to February 24, 2009.
Groups:
- 4 mg/kg: Participants with metastatic non-small-cell lung adenocarcinoma administered 4.0 mg/kg Aflibercept intravenously every 2 weeks until a study withdrawal criterion was met.
Arm/Group | 4 mg/kg
Serious Adverse Events (participants affected / at risk) | 48/96
Other Adverse Events (participants affected / at risk) | 93/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg/kg (N=96)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Obstruction gastric (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Disease progression (General disorders) | 7
Fatigue (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Sepsis (Infections and infestations) | 2
Facial bones fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Radiation injury (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Bladder stenosis (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Axillary vein thrombosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Superior vena caval occlusion (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 4 mg/kg (N=96)
Abdominal pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 27
Diarrhoea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 23
Oral pain (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 16
Chest pain (General disorders) | 5
Disease progression (General disorders) | 6
Fatigue (General disorders) | 39
Mucosal inflammation (General disorders) | 5
Oedema peripheral (General disorders) | 20
Pain (General disorders) | 6
Pyrexia (General disorders) | 11
Pneumonia (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 11
Weight decreased (Investigations) | 9
Anorexia (Metabolism and nutrition disorders) | 24
Decreased appetite (Metabolism and nutrition disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 5
Hyponatraemia (Metabolism and nutrition disorders) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 38
Anxiety (Psychiatric disorders) | 7
Depression (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 10
Proteinuria (Renal and urinary disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 22
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 37
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 8
Hypertension (Vascular disorders) | 38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to independently publish study results from his site after a multicenter publication, or 12 months after the completion of the study by all sites. He must provide the sponsor a copy of any such publication derived from the study for review and comment at least 45 days (20 days for abstracts) in advance of any submission, and delay publication till the approval of the publication is given in writing by the Sponsor (not to exceed ninety days).